CLINICAL TRIAL: NCT00038766
Title: A Randomized, Double-Blind, Placebo-controlled Study of CNI-1493 for Treatment of Moderate to Severe Crohn's Disease
Brief Title: CNI-1493 for Treatment of Moderate to Severe Crohn's Disease
Acronym: CD02
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll into study.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNI-1493 CD-02
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Crohn Disease
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — semapimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Semapimod 60 mg (Experimental): Semapimod 60 mg IV x 5 days
  Interventions: Drug: semapimod
- Semapimod IV 30 mg (Experimental): Semapimod IV 30 mg x 5 days
  Interventions: Drug: semapimod
- Placebo (Placebo Comparator): Placebo IV x 3 or 5 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semapimod — semapipmod 60 mg IV x 5 days
  Other Names: CNI-1493
  Arms: Semapimod 60 mg
Drug: semapimod — IV 30 mg x 5 days
  Other Names: CNI-1493
  Arms: Semapimod IV 30 mg
Drug: placebo — placebo IV
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether CNI-1493 is safe and effective in the treatment of moderate to severe Crohn's Disease.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic inflammatory disease involving the upper and lower gastrointestinal tract and characterized by abdominal pain, weight loss, gastrointestinal bleeding and formation of fistulas between loops of bowel and from the bowel to the skin or other organs. Current therapy for active Crohn's disease consists of symptomatic treatment, nutritional therapy, salicylates and immunosuppressants or surgical management.

Tumor necrosis factor a (TNF-a) plays a central role in the initiation and amplification of the granulomatous inflammatory reaction seen in CD (van Deventer, 1997). Increased TNF-a is present in gut mucosa as well as in stool of patients with active CD (Braegger et al, 1992). CNI-1493 is a synthetic guanylhydrazone compound that is an inhibitor of TNF-a synthesis. A monoclonal antibody to TNF, infliximab, is now approved for treatment of CD, but not all patients respond and many who do respond eventually become refractory to this treatment as well.

CNI-1493 is a synthetic compound which blocks the production of several inflammatory cytokines, including TNF. Because it blocks production of multiple inflammatory mediators, it may be more active than products targeted to a specific cytokine. In addition, as it is not a biologic, it should not cause hypersensitivity reactions or induce formation of antibodies.

The purpose of this trial is to determine if CNI-1493 is safe and effective in treating patients with moderate to severe Crohn's Disease in a placebo controlled setting.

ELIGIBILITY:
Inclusion Criteria

* Baseline Crohn's Disease Activity Index (CDAI) 250-400, inclusive
* Crohn's disease of at least 3 months duration, with colitis, ileitis, or ileocolitis, confirmed by radiography and/or endoscopy
* Patients receiving medications for CD must be on stable doses entering the study
* Any CD medication which has been discontinued must have been discontinued at least 4 weeks prior to screening, with the exception of infliximab, which must have been discontinued at least 8 weeks prior to screening

Exclusion Criteria

* Patients with any ostomy or extensive bowel resection
* Current evidence of bowel obstruction or history within the preceding six months as confirmed by radiography, endoscopy, or surgery
* Patients with stool examination positive for enteric pathogens, pathogenic ova or parasites, or Clostridium difficile toxin
* Treatment with any other experimental therapeutics within the last 4 weeks before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-06; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Change in CDAI | Day 29

SECONDARY OUTCOMES:
Change in IBDQ | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Daan Hommes, M, Principal Investigator — Academic Medical Center, Netherlands
Locations (13):
- United States (13):
  - Institute of Healthcare Assessment, San Diego, California
  - University of Florida, Gainesville, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Long Island Clinical Research Associates, Great Neck, New York
  - Mount Sinai School of Medicine, New York, New York
  - Charlotte Gastroenterology and Hepatology, PLLC, Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - Digestive and Liver Disease Specialists, Norfolk, Virginia

REFERENCES:
- [Background] Hommes D, van den Blink B, Plasse T, Bartelsman J, Xu C, Macpherson B, Tytgat G, Peppelenbosch M, Van Deventer S. Inhibition of stress-activated MAP kinases induces clinical improvement in moderate to severe Crohn's disease. Gastroenterology. 2002 Jan;122(1):7-14. doi: 10.1053/gast.2002.30770. PMID 11781274